CLINICAL TRIAL: NCT00081042
Title: An Open-Label, Multicenter, Phase II Trial of ABI-007 (A Cremophor® -Free, Protein Stabilized, Nanoparticle Paclitaxel) in Previously Treated Patients With Metastatic Melanoma
Brief Title: ABI-007 in Treating Patients With Inoperable Locally Recurrent or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000358804; UCLA-0309060; ABI-CA014
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2005-05

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Taxes

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ABI-007, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well ABI-007 works in treating patients with inoperable (unresectable) locally recurrent or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of ABI-007 in patients with inoperable locally recurrent or metastatic melanoma.
* Determine the safety and tolerability of this drug in these patients.

Secondary

* Determine the time to disease progression, in terms of the rate and duration of response or stable disease, in patients treated with this drug.
* Determine the survival of patients treated with this drug.
* Determine the effects of this drug on biomarkers of melanoma in these patients.
* Correlate biomarker levels with response in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study. Patients are assigned to 1 of 2 treatment cohorts according to prior cytotoxic chemotherapy (previously treated vs chemotherapy-naïve).

* Cohort I (previously treated): Patients receive ABI-007 IV over 30 minutes on days 1, 8, and 15.
* Cohort II (chemotherapy-naïve): Patients receive a higher dose of ABI-007 as in cohort I.

In both cohorts, courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 6 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 24-70 patients (12-35 per cohort) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed melanoma

  * Inoperable locally recurrent or metastatic disease
* Measurable disease

  * No lytic or blastic bone metastasis as only evidence of metastasis
  * Prior radiotherapy to a target lesion allowed provided there has been clear progression of disease since completion of radiotherapy
* No active brain metastasis, including leptomeningeal involvement

  * Prior brain metastasis allowed provided the disease is in complete remission for at least 1 month after therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (unless bone metastasis is present in the absence of liver metastasis)
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception 1 month before and during study participation
* No pre-existing peripheral neuropathy ≥ grade 2
* No prior allergy or hypersensitivity to study drug
* No concurrent clinically significant illness
* No other concurrent active malignancy
* No serious medical risk factors involving any of the major organ systems that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Recovered from prior chemotherapy
* More than 4 weeks since prior cytotoxic chemotherapy
* At least 3 weeks since prior anthracyclines
* No concurrent taxane or anthracyclines
* No concurrent doxorubicin

Endocrine therapy

* No concurrent steroids except as needed for hypersensitivity to study drug

Radiotherapy

* See Disease Characteristics
* Concurrent radiotherapy to a symptomatic non-target lesion (including recurrent or new brain metastases that develop during study participation) allowed

Surgery

* Not specified

Other

* More than 4 weeks since prior investigational drugs and recovered
* No other concurrent anticancer therapy
* No concurrent participation in another clinical study
* No other concurrent investigational therapies
* No concurrent ritonavir, saquinavir, indinavir, or nelfinavir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Hersh EM, O'Day SJ, Ribas A, Samlowski WE, Gordon MS, Shechter DE, Clawson AA, Gonzalez R. A phase 2 clinical trial of nab-paclitaxel in previously treated and chemotherapy-naive patients with metastatic melanoma. Cancer. 2010 Jan 1;116(1):155-63. doi: 10.1002/cncr.24720. PMID 19877111